CLINICAL TRIAL: NCT02787590
Title: Simvastatin as a Neuroprotective Treatment for Parkinson's Disease: a Double-blind, Randomised, Placebo Controlled Futility Study in Patients of Moderate Severity.
Brief Title: Simvastatin as a Neuroprotective Treatment for Moderate Parkinson's Disease
Acronym: PD STAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Collaborators: University of Plymouth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDSTAT2015; 2015-000148-40 (EudraCT Number); 16108482 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
Keywords: Neurology
MeSH Terms: conditions — Parkinson Disease | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): A one month low dose phase of 40mg oral simvastatin daily will be followed by a 23 month high dose phase of 80mg oral simvastatin daily and a final two month phase off trial medication
  Interventions: Drug: Simvastatin
- Matched Placebo (Placebo Comparator): A one month low dose phase of 40mg matched placebo daily will be followed by a 23 month high dose phase of 80mg matched placebo daily and a final two month phase off trial medication
  Interventions: Drug: Matched Placebo (for Simvastatin)

INTERVENTIONS:
Drug: Simvastatin
  Arms: Simvastatin
Drug: Matched Placebo (for Simvastatin)
  Arms: Matched Placebo

SUMMARY:
Participants are randomly allocated to one of two treatment groups. In one group, participants are given capsules of simvastatin to take orally (by mouth) for 24 months. In the other group, participants are given placebo (dummy) capsules to take orally for 24 months. At the start of the study, when they receive their medication, participants complete a number of questionnaires and motor (movement) tests (a walking test and a finger tapping test). Participants in both groups also attend a further 6 clinic visits after 1, 6, 12, 18 and 24 and 26 months, where they are asked about their health and any medication they are taking, as well as repeating the questionnaires and motor tests. For 4 of the clinic visits, the participants will be asked to attend in the 'OFF medication' state (having omitted their usual PD medication) so that the researchers can get a true picture of their disease without it being masked by their normal medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* Modified Hoehn and Yahr stage ≤ 3.0 in the ON medication state
* Age 40-90 years
* On dopaminergic treatment with wearing-off phenomenon
* Able to comply with study protocol and willing to attend necessary study visits

Exclusion Criteria:

* Diagnosis or suspicion of other cause for parkinsonism
* Known abnormality on CT or MRI brain imaging considered to be causing symptoms or signs of neurological dysfunction, or considered likely to compromise compliance with study protocol
* Concurrent dementia defined by MoCA score <21
* Concurrent severe depression defined by MADRS score >31
* Prior intracerebral surgical intervention for PD including deep brain stimulation, lesional surgery, growth factor administration, gene therapy or cell transplantation
* Already actively participating in a research study that might conflict with this trial
* Prior or current use of statins as a lipid lowering therapy
* Intolerance to statins
* Untreated hypothyroidism
* End stage renal disease (creatinine clearance <30 mL/min) or history of severe cardiac disease (angina, myocardial infarction or cardiac surgery in preceding two years)
* eGFR <30 mL/min
* History of alcoholism or liver impairment
* Creatine kinase (CK) >1.1 x upper limit of normal (ULN)
* Aspartate transaminase (AST) or alanine transaminase (ALT) >1.1 x ULN
* Females who are pregnant or breast feeding or of child-bearing potential and unwilling to use appropriate contraception methods whilst on trial treatment
* Currently taking any medication contraindicated with simvastatin use (Appendix 2)
* Any requirement for statin use
* Regular participation in endurance or high-impact sports
* Unable to abstain from consumption of grapefruit-based products

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in MDS-UPDRS part III (OFF) score | Baseline and 24 Months
  The MDS-UPDRS is the standard validated tool for the assessment of patients with Parkinson's Disease. This scale includes subsections collecting data regarding the impact of PD on a patient's mood and mental state, (UPDRS part I), their activities of daily living (UPDRS part II) an examination of the motor features of PD (UPDRS part III), and complications arising from the use of dopamine replacement (part IV).

SECONDARY OUTCOMES:
MDS-UPDRS total score in the practically defined ON state | at 12 and 24 months
MDS-UPDRS part II subscale score in the practically defined ON state | at 12 and 24 months
Timed motor tests - finger tapping and timed walk test (10MWT) in the OFF state, electromagnetic sensor (EMS) assessment in the OFF and ON state | at 12 and 24 months
  Timed Motor Tests include evaluating the number of hand taps (key strokes) that an individual can perform within 30 seconds and a timed walk test (10MWT). Electromagnetic Sensor Measurements include wearing sensors on the index finger and thumb whilst performing 4 MDS-UPDRS items.
Montgomery and Asberg Depression Rating Scale (MADRS) | at 12 and 24 months
  The Montgomery and Asberg Depression Rating Scale (MADRS) is a 10 item physician rated depression severity scale previously used in the assessment of PD
The Addenbrooke's Cognitive Assessment-III (ACE-III) | at 12 and 24 months
  The Addenbrooke's Cognitive Examination-III (ACE) is one of the most popular and PD STAT protocol version 2.2, 03 March 2016 EudraCT 2015-000148-40 ISRCTN16108482. REC Ref:15/NE/0324 Page 39 of 43 commonly used cognitive tests used in dementia clinics and in the assessment of other neurological disorders. ACE-III includes five subdomains which provide a cognitive score out of a maximum of 100
Non-Motor Symptom assessment scale (NMSS) | at 12 and 24 months
  The Non-Motor Symptom assessment scale (NMSS) is a rating scale designed to capture the presence of the non-motor features of PD
Parkinson's disease Questionnaire (PDQ-39) | at 12 and 24 months
  The PDQ39 is a PD-specific health status questionnaire used both clinically and within research since its publication in 1995. It consists of 39 items covering eight discrete dimensions: mobility, emotional well-being, stigma, social support, cognition, communication and bodily discomfort. The scores from each dimension are computed into a scale ranging from 0 (best, i.e. no problem at all) to 100 (worst, i.e. maximum level of problem). In addition a summary score, the PDQ-39SI (summary index) can be calculated by averaging the scores of the eight dimensions.
Changes in PD medication as measured by levodopa-equivalent dose (LED) | at 12 and 24 months
Cholesterol levels (total, HDL, total/HDL ratio) | at 12 and 24 months
King's PD pain scale (KPPS) | at 12 and 24 months
  The King's PD Pain Scale is a PD-specific scale consisting of 14 items within seven domains. Each item is scored by severity (0-3) multiplied by frequency (0-4), resulting in an item sub-score of 0-12 and a total possible score of 0-168.
EuroQoL 5D-5L health status questionnaire (EQ-5D-5L) | at 12 and 24 months
Safety and tolerability of trial medication by adverse events (AEs) review. | at 12 and 24 months
Incidence of diabetes mellitus, using a glycated haemoglobin (HbA1c) level of 6.5% (48mmol/mol) as diagnostic of diabetes mellitus. | at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Camille B Carroll, BM BCh, PhD, Study Director — Clinical Lecturer (University of Plymouth) and Honorary Consultant Neurologist, Plymouth Hospitals NHS Trust.
Locations (24):
- United Kingdom (24):
  - Royal United Hospital, Bath
  - Royal Bournemouth Hospital, Bournemouth
  - Fairfield General Hospital, Bury
  - Addenbrooke's Hospital, Cambridge
  - St Peter's Hospital, Chertsey
  - Royal Devon and Exeter Hospital, Exeter
  - Leeds General Infirmary, Leeds
  - Charing Cross Hospital, London
  - King's College Hospital, London
  - Royal Free Hospital, London
  - Luton and Dunstable Hospital, Luton
  - Clinical Ageing Research Unit, Newcastle
  - Norfolk and Norwich University Hospital, Norwich
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Queen's Hospital, Romford
  - Rotherham General Hospital, Rotherham
  - Salford Royal Hospital, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Musgrove Park Hospital, Taunton
  - Royal Cornwall Hospital, Truro
  - Yeovil District Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plans for the current study are unknown and will be made available at a later date
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: On application

REFERENCES:
- [Derived] Carroll CB, Webb D, Stevens KN, Vickery J, Eyre V, Ball S, Wyse R, Webber M, Foggo A, Zajicek J, Whone A, Creanor S. Simvastatin as a neuroprotective treatment for Parkinson's disease (PD STAT): protocol for a double-blind, randomised, placebo-controlled futility study. BMJ Open. 2019 Oct 7;9(10):e029740. doi: 10.1136/bmjopen-2019-029740. PMID 31594876
- See also: Trial website — https://penctu.psmd.plymouth.ac.uk/pdstat/Default.aspx